CLINICAL TRIAL: NCT06731725
Title: Post-marketing Study to Evaluate the Efficacy of I+MED's DayDrop in Improving Mild/Moderate Dry Eye Symptoms
Brief Title: Post-marketing Study Focused on Evaluating I+Med's DayDrop for Improving Signs and Symptoms of Mild/Moderate Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Bioaraba Health Research Institute (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DayDrop-PIC01-2020
Record Dates: First submitted 2024-12-04; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye; Dry Eye Syndrome (DES)
Keywords: Dry eye; DayDrop; Opthalmic Tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Clinical post-marketing quasi-experimental before-and-after trial, which includes 20 patients diagnosed with mild/moderate dry eye disease (defined by a score on the OSDI test ≥13 and ≤22) who attend the ophthalmology consultation at the outpatient building of the Araba University Hospital and meet the inclusion criteria with no exclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DayDrop® (Experimental): Medical Device IIa class. DayDrop is a biocompatible ophthalmic solution indicated to relieve dryness and ocular irritation. DayDrop is composed of ectoine, carboxymethylcellulose, and sodium hyaluronate. The product is obtained by dissolving the components in a borate buffer (pH = 7.2-7.6) prepared with boric acid and sodium tetraborate. The manufacturing and packaging of the product are carried out under aseptic processing conditions following the UNE-EN ISO 13408:2015 standard, and the product is sterilized through sterilizing filtration. DayDrop is defined as a sterile product, buffered to a neutral pH, phosphate-free, preservative-free, and compatible with contact lenses according to ISO 11981.
  Interventions: Device: DayDrop®

INTERVENTIONS:
Device: DayDrop® — The patient will administer 1 to 2 instillations each time it is necessary (at least 2 times a day) and will record it in their data collection notebook.

SUMMARY:
Clinical post-marketing quasi-experimental before-and-after trial to determine the effectiveness of DayDrop treatment in subjects seeking relief from symptoms of dryness and eye irritation based on OSDI questionnaire scores completed by patients.The study will involve 20 patients diagnosed with mild/moderate dry eye disease who meet the inclusion/exclusion criteria. The duration of the study will be 2 weeks, including 3 visits.

DETAILED DESCRIPTION:
Clinical post-marketing quasi-experimental before-and-after trial to determine the effectiveness of DayDrop treatment in subjects seeking relief from the signs of dryness and eye irritation, comparing the scores obtained at the end of the follow-up period with those established before the start of treatment (baseline condition), as measured by the patients according to the OSDI questionnaire.

The study will involve 20 patients diagnosed with mild/moderate dry eye disease who meet the inclusion/exclusion criteria of the protocol. The study duration will be 2 weeks, including 3 visits: baseline, visit 1 (after one week of treatment), and visit 2 (at 2 weeks from the start of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over 18 years of age.
* Patients presenting symptoms of dryness and ocular irritation with an OSDI score ≥13 and ≤22.
* Ability to self-administer the drops.
* Ability to understand the Patient Information Sheet and sign the Informed Consent.
* Willingness and sufficient ability, as judged by the investigator, to respond to the questionnaires included in the study.

Exclusion Criteria:

* Pregnant women or those in the breastfeeding period.
* Known allergy or hypersensitivity to hyaluronic acid or any other ingredient in the product being studied.
* Patients who have undergone previous ocular surgery or experienced ocular trauma in the year prior to the start of the study.
* Severe dry eye diagnosis.
* Presence of inflammatory ocular surface pathology or anterior segment disease, or diagnosed with glaucoma.
* Use of parasympathomimetic or antipsychotic medications.
* Previous cataract surgery.
* Systemic corticosteroid treatment or topical treatment with any ophthalmic medication, except artificial tears, in the week before the start of the study.
* Sjögren's syndrome.
* Stevens-Johnson syndrome.
* History of allergic conjunctivitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Change in the score obtained in the OSDI questionnaire. | At baseline and in week 3
  The OSDI questionnaire will be completed by the patients and is used to analyze the presence of progress in dry eye symptoms. The 12 questions of the OSDI questionnaire will be used to calculate the index (total score range from 0 to 48). The score obtained for these parameters at the start of the study (baseline) will be compared with the score obtained at the end of the follow-up period.
  To support the hypothesis of effectiveness, treatment with DayDrop will result in a significant improvement (of at least 6 points out of 48) in the OSDI index scores at the end of the follow-up period, compared to the values recorded at the start of the study.

SECONDARY OUTCOMES:
Change in the score obtained in the OSDI questionnaire at week 1. | At week 1
  he 12 questions of the OSDI questionnaire will be used to calculate the index (total score range from 0 to 48). The score obtained for these parameters at the start of the study (baseline) will be compared with the score obtained at the end of the follow-up period.
  To support the hypothesis of effectiveness, treatment with DayDrop will result in a significant improvement (of at least 6 points out of 48) in the OSDI index scores at the end of the follow-up period, compared to the values recorded at the start of the study.
Assessment by the investigators of the treatment's effectiveness. | At week 2
  A questionnaire for the final evaluation of the treatment will be provided to the investigator. A questionnaire for the final evaluation of the treatment will be provided to the investigator. A response rate will be calculated, which should be at least 50% of responders, defined as those cases rated as "Improvement," "Significant Improvement," or "Exceptional Improvement."
Evaluation by the subjects of the treatment's effectiveness. | At week 2
  A questionnaire for the final evaluation of the treatment will be provided to the patients. In an exploratory manner, global improvement in terms of the frequency and severity of symptoms will be assessed at the end of the treatment. A satisfaction rating of "Satisfied," "Very Satisfied," or "Exceptionally Satisfied" is expected in at least 50% of the cases. Additionally, the duration of the effect and the number of times drops were needed will be evaluated in comparison to other eye drops previously used (≥ 50% of patients rating the effect as at least as long-lasting and using the same or fewer daily drops compared to other eye drops used previously).
Adverse events. | Through study completion, apprroximately 3 weeks
  Evaluating number and severity of adverse events through the systematic recording and analysis of the events and incidents detected during the study. The incidence of incidents with DayDrop should be significantly low and should not exceed the threshold set at 1%.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Álava, Spain